CLINICAL TRIAL: NCT03642236
Title: Combination of Brutons Tyrosine Kinase (BTK) Inhibitor Overcomes Drug-resistance in Refractory/Relapsed FLT3 Mutant Acute Myeloid Leukemia (AML)
Brief Title: Combination of BTK Inhibitor Overcomes Drug-resistance in Refractory/Relapsed FLT3 Mutant AML
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, yuguopan, professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTKi in FLT3 mutant AML
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: FLT3-ITD Mutation; Acute Myeloid Leukemia; Brutons Tyrosine Kinase
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BTK treatment (Experimental): Ibrutinib 420mg day -3 to d14; Decitabine 20mg/m2 d1-5; Aclacinomycin 10mg/m2 d1-5; Cytarabine 15mg/m2 q12h d1-14; G-CSF 200ug/m2 -12h to d14; Sorafenib 0.4g bid continously at the condition of being naive to sorafenib.
  Interventions: Drug: Ibrutinib
- BTK-free treatment (Active Comparator): Decitabine 20mg/m2 d1-5; Aclacinomycin 10mg/m2 d1-5; Cytarabine 15mg/m2 q12h d1-14; G-CSF 200ug/m2 -12h to d14; Sorafenib 0.4g bid continously at the condition of being naive to sorafenib.
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib 420mg day -3 to d14 combining with chemotherapy with/without sorafenib based on whether the patients are naive to sorafenib before relapse.

SUMMARY:
Clinical efficacy of FLT3 inhibitors combining with chemotherapy is usually transient and followed by emergence of drug-resistance in FLT3-ITD mutant AML. BTK is reported to be a therapeutic target in this subtype leukemia. Our previous study showed inhibition of BTK onvercome drug-resistance to FLT3 inhibitors/chemotherapy in refractory/relapsed FLT3 mutant AML. In this prospective randomized controlled study, the efficacy and safety of combination of BTK inhibitor with chemotherapy with/without FLT3 inhibitor in refractory/relapsed FLT3 mutant AML are evaluated.

DETAILED DESCRIPTION:
Clinical efficacy of FLT3 inhibitors combining with chemotherapy is usually transient and followed by emergence of drug-resistance in FLT3-ITD mutant acute myeloid leukemia (AML). How to overcome the resistance to FLT3 inhibitors or chemotherapy needs further study. Bruton's tyrosine kinase (BTK) is reported to be a therapeutic target in this subtype leukemia. Our previous study showed inhibition of BTK onvercome drug-resistance to FLT3 inhibitors/chemotherapy in refractory/relapsed FLT3 mutant AML. In this prospective randomized controlled study, we are going to inhibit BTK with BTK inhibitor ibrutinib in the patients with refractory/relapsed FLT3 mutant AML, and then test the enhancing effect and safety of combination of ibrutinib with chemotherapy with/without FLT3 inhibitor, to make sure inhibition of BTK overcomes drug-resistance in FLT3 mutation AML.

ELIGIBILITY:
Inclusion Criteria:

Refractoty/relapsed FLT3-ITD mutation AML Age 14-60

Exclusion Criteria:

Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure) Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 122 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
CR rate | After the first and second cycle induction
OS | 2 years
DFS | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Guopan Yu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China